CLINICAL TRIAL: NCT06452017
Title: Effects of Telerehabilitation Exercise Program on Maternal Antenatal Glycemic Control in Women With Gestational Diabetes.
Brief Title: Effects of Telerehabilitation Exercise Program on Maternal Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Maheen Haq
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Intervention Model Description: there will be comparison between the two groups, experimental and control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telerehabilitation exercise group (Experimental): this group will receive a structured telerehabilitation exercise protocol of low to moderate intensity warm up ,aerobic ,resistance and cool down exercises for 3 times a week progressively increased for 8 weeks in addition to routine medical care for GDM.
  Interventions: Other: Telerehabilitation exercise program
- routine medical care (Active Comparator): The control group will receive routine medical care including oral medication,diet and regular walk.
  Interventions: Other: Routine medical care

INTERVENTIONS:
Other: Telerehabilitation exercise program — 5 min warmup will include ankle plantar and dorsiflexion ,trunk side flexion ,shoulder circles ,shoulder ROMS.it will be followed by 5 min aerobics that includes spot marching and side stepping. it will be followed by resistance exercise which will be divided into 3 groups. each group of exercise will be performed one day each. chair squats, arm pulls, seated triceps, biceps curls etc. are included in these resistance exercises. intensity of each exercise will be progressively increased.
  Arms: telerehabilitation exercise group
Other: Routine medical care — The control group will be given routine medical care (including dietary modification, oral anti diabetics (metformin) and advised to do regular walk (20-30min/day).
  Arms: routine medical care

SUMMARY:
Gestational diabetes is in which high blood glucose concentration results from body's inability to create enough insulin to fulfil the needs of pregnancy. It appears in week between 24 to 28 and and raises the mothers and Childs risk of problems. It is thought to affect about 1 in 7 pregnancies worldwide. Through these remote exercise sessions the study evaluates the effectiveness of tele rehabilitation in improving glycemic management during pregnancy.The results will help clarify how telehealth intervention can best support GDM patient's maternal health outcomes.

DETAILED DESCRIPTION:
Literature suggests that hormonal changes during pregnancy can interfere with insulin, the hormone that regulates blood glucose.This excess glucose can cross the placenta, affecting the developing fetus and increasing risks for both mother and child. The rising trends in obesity and advanced maternal age suggest that the prevalence of GDM will continue to increase.Approximately 7-10% of pregnancies worldwide are affected by gestational diabetes.Managing glucose levels is critical for women with gestational diabetes to ensure a healthy pregnancy and reduce the risk of complications for both mother and baby. Developing a positive attitude towards exercise is important for helping people with gestational diabetes manage their condition effectively through physical activity. The use of telerehabilitation may improve blood glucose levels in participants with GDM.

The control group will receive routine medical care and the experimental group will receive structured telerehabilitation exercise protocol. The results of both groups will be recorded and compared to assess the effectiveness of using telerehabilitation in the treatment of women with GDM in improving maternal blood glucose level.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 to 35 years
* Gestational age between 20-28weeks
* diagnosed with Gestational diabetes mellitus through oral glucose tolerance test (OGTT)
* Primigravida and multigravida
* able to do 6 6-minute walk tests under a severity level of 6 on the Borg scale of breathlessness.
* Patients or caregivers have and able to use an electronic device (PC, tablet or smartphone)
* Who signed informed consent

Exclusion Criteria:

* Previously diagnosed T1DM or T2DM
* High-risk pregnancy conditions contraindicating exercise as per ACOG guidelines
* Patients taking insulin regularly.
* Patients with fetal anomalies diagnosed at 20 th week.
* Multiple gestation (twin or triplets)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Blood sugar fasting | Baseline to 2nd,4th,6th and 8th week
  It is a diagnostic tool to assess person bloods sugar control and screen for diabetes and pre diabetes, is a fundamental measure of blood glucose levels in a fasting state, typically measured after an overnight fast. It provides insights into a person's current blood sugar status and is often used for diagnosing and monitoring diabetes.
Blood sugar random | Baseline to 2nd,4th,6th and 8th week
  Random blood sugar, is a fundamental measure of blood glucose levels after a meal, it will be done 2 hours postprandial.
HbA1c: Glycated hemoglobin | Baseline to 12th week
  This test provides an estimate over average blood glucose level over past two to three months. It is a critical clinical marker used to assess long-term blood sugar control in individuals with diabetes. It measures the percentage of hemoglobin in the blood that has glucose attached to it.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PhD, Principal Investigator — Riphah International University, Islamabad, Pakistan
Locations (2):
- Pakistan (2):
  - Pakistan Railway hospital, Rawalpindi, Punjab Province
  - AlKhidmat Razi Hospital,Rawalpindi, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munoz-Tomas MT, Burillo-Lafuente M, Vicente-Parra A, Sanz-Rubio MC, Suarez-Serrano C, Marcen-Roman Y, Franco-Sierra MA. Telerehabilitation as a Therapeutic Exercise Tool versus Face-to-Face Physiotherapy: A Systematic Review. Int J Environ Res Public Health. 2023 Feb 28;20(5):4358. doi: 10.3390/ijerph20054358. PMID 36901375
- [Background] Bung P, Artal R, Khodiguian N. [Regular exercise therapy in disorders of carbohydrate metabolism in pregnancy--results of a prospective, randomized longitudinal study]. Geburtshilfe Frauenheilkd. 1993 Mar;53(3):188-93. doi: 10.1055/s-2007-1023663. German. PMID 8467987
- [Background] Stafne SN, Salvesen KA, Romundstad PR, Eggebo TM, Carlsen SM, Morkved S. Regular exercise during pregnancy to prevent gestational diabetes: a randomized controlled trial. Obstet Gynecol. 2012 Jan;119(1):29-36. doi: 10.1097/AOG.0b013e3182393f86. PMID 22183208
- [Background] Tobias DK, Zhang C, van Dam RM, Bowers K, Hu FB. Physical activity before and during pregnancy and risk of gestational diabetes mellitus: a meta-analysis. Diabetes Care. 2011 Jan;34(1):223-9. doi: 10.2337/dc10-1368. Epub 2010 Sep 27. PMID 20876206